CLINICAL TRIAL: NCT00056901
Title: A Screening Protocol to Evaluate Women With Postpartum-Related Mood and Behavioral Disorders
Brief Title: Screening Evaluation for Women With Postpartum Depression
Status: Terminated | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030138; 03-M-0138
Record Dates: First submitted 2003-03-26; First posted 2003-03-26 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2017-12-24

CONDITIONS: Postpartum Depression; Depression
Keywords: Puerperium; Pregnancy; Mood Disorders; Estradiol; Progesterone; Mood; Behavior; Cognition; Perimenopause; Menopause; Post Partum Depression; PPD; Healthy Volunteer; HV
MeSH Terms: conditions — Depression, Postpartum; Depression; Mood Disorders; Behavior

SUMMARY:
This study evaluates the relationship between mood changes and hormones in women with postpartum depression (PPD).

This is an observational study; volunteers who participate will not receive any new or experimental therapies.

PPD is similar to major depression, but develops around the time a woman gives birth. Women with PPD often suffer serious physical and emotional impairments. Controversy exists regarding the role of hormone changes in postpartum depression. This study will examine the role of hormone changes in three groups of women: those who recently gave birth and have mild to moderately severe PDD (Group 1), women who recently gave birth and do not have PDD (Group 2), and those who are currently pregnant and experienced an episode of PDD with a previous birth (Group 3).

Participants will be screened with a medical history, physical examination, and blood and urine tests. Upon study entry, they will be interviewed about their moods, behaviors, and medical status during and immediately following their last pregnancy. Some women will be asked to participate in interviews, psychological tests, and blood tests. They will also complete self-rating scales and may be asked to collect samples of their urine. Women in Group 3 will complete self-rating scales for 6 months postpartum. Participants will participate in genetic studies that involve completing a questionnaire and providing a blood sample. If the participant allows, sisters and parents may be asked to provide a blood sample and undergo a psychiatric interview.

Participants who meet the criteria for minor depression or major depression that is no greater than moderate severity will be asked to participate in a companion study that will evaluate the effectiveness of estradiol in reducing depression symptoms.

...

DETAILED DESCRIPTION:
Controversy exists regarding the relevance of changes in gonadal steroids for postpartum-onset depressions. The purpose of this protocol is to allow for the careful screening of patients and healthy volunteers for participation in research protocols that examine the role of gonadal steroids in postpartum-onset depressions (PPD) and for the collection of natural history data. Women in this protocol will undergo an evaluation which may include: a psychiatric interview; a diagnostic interview; rating scales; a medical history; a physical exam; blood and urine laboratory evaluation; and a request for medical records. The data collected may also be linked with data from other PPD protocols (e.g., DNA, psychophysiology tests, treatment studies, etc.) for the purposes of better understanding the diagnosis, pathophysiology, and treatment response of women with PPD. Upon conclusion of the screening process, subjects will either be offered participation in a research protocol and will sign the appropriate informed consent, or will be considered not appropriate for participation in research and will be referred back into the community. The second purpose of this protocol is to permit the identification of pregnant women who are at risk for developing postpartum depression (PPD), and who are followed longitudinally through the postpartum in an effort to confirm the association of depression onset with change in reproductive endocrine function. This protocol, then, serves as a screening and evaluation protocol to recruit subjects who are characterized with standard measures in this protocol and then offered participation in related studies.

ELIGIBILITY:
* INCLUSION CRITERIA:

Cross-sectional Screening: The postpartum subjects of this protocol will be women who meet the following inclusion criteria:

* History of at least two weeks with postpartum-related mood or behavioral disturbances of at least moderate severity - that is, disturbances that are distinct in appearance and associated with a mild to moderate degree of functional impairment;
* The onset of mood symptoms occurred within three months of delivery;
* Age 20-45; The selection of the lower limit of this age window is intended to reduce the potential confound that the psychosocial stress of a teenage pregnancy could complicate the relationship between postpartum hormonal events and mood. The upper age limit was selected since pregnancy and childbirth in a woman over this age range could lead to spontaneous menopause and, therefore, our ability to discern the effects of estrogen therapy on mood could be complicated by estrogen s effects on menopausal symptoms.
* History of normal delivery (vaginal or caesarean) within last six months;
* No prior estrogen replacement therapy for treatment of postpartum physical or emotional symptoms within the last six months;
* In good medical health.
* Subjects must be competent to comprehend the purpose of the screening process and to provide written informed consent and be willing to participate in NIMH IRB approved research protocols.
* A control group of age-matched postpartum women who meet patient selection criteria with the exception of the presence of mood or behavioral disorders will also be sought.

EXCLUSION CRITERIA:

* Current antidepressant therapy
* Subjects should have no general medical illness that is primary (i.e., appears to be causing the mood disorder);
* Current alcohol or substance use or dependence (excluding nicotine) of sufficient magnitude to require independent, concurrent treatment intervention (e.g., antabuse or opiate treatment, but not including self-help groups).
* This protocol is a screening protocol for an estradiol treatment study (03-M-0161) for which the exclusion criteria include the current use of antidepressant medications. However, antidepressants will not be withheld from subjects who need or want them. Immediately after screening subjects will either be enrolled in the estrogen treatment study or in traditional therapy until care can be transitioned to the community. There are few exclusion criteria for the evaluation component of this protocol; however, all women will undergo a structured diagnostic interview Those women who will be asked to participate in the companion protocol evaluating the efficacy of estradiol administration in PPD will meet either research diagnostic criteria for minor depression with at least three core symptoms (SADS-L (90) or major depression (SCID-IV) (91) of not greater than moderate severity on the Global Assessment of Functioning Scale (GAF) (91)) and will not meet DSM-IV criteria # 9 (suicide) or require immediate treatment. Subjects meeting major depression with greater than moderate severity may participate in the evaluation phase of this study but will be offered a referral to an outside facility for standard antidepressant treatment (i.e., they are not candidates for participation in the IRB approved treatment protocol).

LONGITUDINAL SCREENING:

INCLUSION CRITERIA FOR THE AT RISK PREGNANT WOMEN:

* Pregnant;
* Absence of current mood or behavioral disturbance as determined by a structured diagnostic interview;
* Past history of postpartum depression;
* In good medical health,
* Medication free.

GENETIC STUDIES:

INCLUSION CRITERIA:

Unaffected family members of women with PPD will be admitted for genetic studies only who are first degree relatives of women with confirmed PPD, and who do not have PPD as defined in this protocol.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2003-03-25; Study Completion 2017-12-24

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Schmidt, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kumar R, Robson KM. A prospective study of emotional disorders in childbearing women. Br J Psychiatry. 1984 Jan;144:35-47. doi: 10.1192/bjp.144.1.35. PMID 6692075
- [Background] Cox JL, Murray D, Chapman G. A controlled study of the onset, duration and prevalence of postnatal depression. Br J Psychiatry. 1993 Jul;163:27-31. doi: 10.1192/bjp.163.1.27. PMID 8353695
- [Background] O'Hara MW, Schlechte JA, Lewis DA, Varner MW. Controlled prospective study of postpartum mood disorders: psychological, environmental, and hormonal variables. J Abnorm Psychol. 1991 Feb;100(1):63-73. doi: 10.1037//0021-843x.100.1.63. PMID 2005273